CLINICAL TRIAL: NCT04714775
Title: Validation of Biomarkers of Adverse Neurologic Outcome in Newborns at Risk for Perinatal Brain Injury - Study on Neuro-developmental Follow-up at 2 Years A Prospective Multicenter Observational Study for Development of a Diagnostic Test
Brief Title: Biomarkers And Neurological Outcome in Neonates 2
Acronym: BANON2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: InfanDx AG (Industry)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: BANON2
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Asphyxia Neonatorum
Keywords: Biomarkers; Asphyxia; Hypoxic ischemic encephalopathy
MeSH Terms: conditions — Asphyxia Neonatorum; Asphyxia; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Follow-up of participants of BANON1 study at age of at least 2 years. BANON1 (ClinicalTrials.gov ID: NCT03357250): Validation of biomarkers based on 24 months neuro-developmental outcome data in a human population for their ability to diagnose the severity of neonatal asphyxia. These biomarkers linked to asphyxia have been identified in animal studies and a preliminary human study.

DETAILED DESCRIPTION:
Follow-Up on neuro-developmental status of Study participants of BANON1. BANON1 (ClinicalTrials.gov ID: NCT03357250): The aim of the study is to validate the application of combinations of several laboratory parameters in early postnatal blood samples, for identification of infants, who will suffer from early abnormal neonatal neurological outcome, in a population at risk. The population at risk is defined as term and late preterm (>36 weeks of gestation) human infants following perinatal hypoxia-ischemia with or without postnatal resuscitation, and where the combination of laboratory parameters is derived from a preliminary study performed in Turkey (AAMBI) using a metabolomics approach.

ELIGIBILITY:
Inclusion Criteria:

* Infants previously enrolled in BANON study

Exclusion Criteria:

* Missing valid written informed parental consent

Ages: 22 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, who had been enrolled in the BANON study immediately after birth because they had been suspected to be at risk for perinatal brain injury (hypoxic-ischemic encephalopathy, HIE) and/or evaluated for hypothermia therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
participants with normal neuro-developmental status | up to 42 month age
  all infants with normal neuro-developmental status
participants with potentially abnormal neuro-developmental status | up to 42 month age
  All infants who do not fulfill outcomes 1, 3 or 4
participants with abnormal neuro-developmental status - HIE | up to 42 month age
  Presence of adverse 2 years neuro-developmental outcome likely attributable to perinatal hypoxic-ischemic brain injury
participants with abnormal neuro-developmental status - non-HIE | up to 42 month age
  Presence of adverse 2 years neuro-developmental outcome not attributable to perinatal hypoxic-ischemic brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Ron Meyer, Study Director — InfanDx AG
Locations (13):
- Germany (11):
  - Städtisches Krankenhaus Aschaffenburg, Aschaffenburg
  - Universitätsklinikum Carl Gustav Carus, Neonatologie, Dresden
  - Uniklinik Essen, Essen
  - Marienkrankenhaus, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Städtisches Klinikum Karlsruhe, Klinik für Kinder- und Jugendmedizin, Karlsruhe
  - Klinik für Kinder- und Jugendmedizin, Klinikum Dritter Orden,, München
  - Universitäts Kinderkrankenhaus und Perinatal Zentrum, München
  - Kinderklinik Dritter Orden, Passau
  - Klinik St. Hedwig, Regensburg
  - Universitätsklinikum Tübingen, Universiätsklinik für Kinder- u. Jugendmedizin, Tübingen
- Turkey (Türkiye) (2):
  - Cukurova University Hospital, Adana
  - University of Firat, Department of Pediatrics, Elâzığ